CLINICAL TRIAL: NCT02509923
Title: A Randomized, Open-label, Crossover, Pharmacokinetic and Pharmacodynamic Study of Z-215 Compared With Rabeprazole Sodium in Healthy Male Subjects
Brief Title: To Evaluate Pharmacokinetics and Pharmacodynamics of Z-215 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Z215-02
Record Dates: First submitted 2015-07-21; First posted 2015-07-28 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: Male Subjects
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 3-way cross-over, Z-215 10 mg/day / Z-215 20 mg/day / Rabeprazole Sodium 10 mg/day
  Interventions: Drug: Z-215 10mg; Drug: Z-215 20mg; Drug: Rabeprazole Sodium 10mg
- 2 (Experimental): 3-way cross-over, Z-215 20 mg/day / Z-215 40 mg/day / Rabeprazole Sodium 20 mg/day
  Interventions: Drug: Z-215 20mg; Drug: Rabeprazole Sodium 20mg
- 3 (Experimental): 3-way cross-over, Z-215 20 mg/day (before breakfast) / Z-215 20 mg/day (after breakfast) / Rabeprazole Sodium 10 mg/day (after breakfast)
  Interventions: Drug: Z-215 20mg; Drug: Rabeprazole Sodium 10mg

INTERVENTIONS:
Drug: Z-215 10mg — Z-215 10mg, capsules
  Arms: 1
Drug: Z-215 20mg — Z-215 20mg, capsules
Drug: Rabeprazole Sodium 10mg — Rabeprazole Sodium 10mg tablets
  Arms: 1; 3
Drug: Rabeprazole Sodium 20mg — Rabeprazole Sodium 20mg tablets
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics and pharmacodynamics of Z-215 (10 mg, 20 mg, 40 mg) , compared with Rabeprazole Sodium (10 mg, 20 mg ) in Healthy Male Subjects. And to evaluate food-effect in Healthy Male Subjects administrated Z-215 20 mg.

ELIGIBILITY:
Inclusion Criteria:

* Has negative results for H. pylori IgG antibody at screening.
* A body mass index 18.5≦BMI<25.0 kg/m^2 at screening.
* Able to understand the consent of the study and comply with the study. Able to give informed consent in writing before participating in the study.

Exclusion Criteria:

* Has a history of PPI allergy.
* Has a history of drug or food serious allergy.
* Presently has or has a history of diseases that may affect evaluation of the study results such as gastrointestinal, hepatic, renal, respiratory, endocrine, blood, cardiovascular, mental or congenial metabolic disease.
* Has a history of surgery (such as resection of the liver, kidney, or digestive tract) that may affect the pharmacokinetics of the study drug.
* History of previous and current acid-related diseases.
* Received H. pylori eradication treatment within 6 months before screening.
* Has 450msec<QTC by Fridericia test at screening ECG .
* Has hypoacidity or anacidity. Or be determined that low gastric acid or no stomach acid by the gastric pH monitoring at baseline period.
* History or suspicion of drug, opioid, alcohol abuse or positive screening results.
* Use of any prescription drugs within 4 weeks prior to baseline period.
* Use of any over-the-counter drugs within 2 weeks prior to baseline period.
* Received blood transfusions within 12 weeks or donated ≥400mL of whole blood within 12 weeks or ≥200mL of whole blood within 4 weeks prior to baseline period. Donated platelet or plasma within 2 weeks prior to baseline period.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
24-Hour Intragastric pH Profile | 4 weeks
  Summary statistics of the measurements on Day1 and Day5 of administration are to be calculated by dose.
Cmax: Maximum Plasma Concentration for Z-215 | 4 weeks
  Summary statistics of pharmacokinetic parameters on Day1 and Day5 of administration are to be calculated by dose.
tmax: Time to Reach Maximum Plasma Concentration (Cmax) for Z-215 | 4 weeks
  Summary statistics of pharmacokinetic parameters on Day1 and Day5 of administration are to be calculated by dose.
t1/2: Terminal Elimination Half-life (t1/2) for Z-215 | 4 weeks
  Summary statistics of pharmacokinetic parameters on Day1 and Day5 of administration are to be calculated by dose.
Lambda Z: Terminal Elimination Rate Constant (Lambda Z) for Z-215 | 4 weeks
  Summary statistics of pharmacokinetic parameters on Day1 and Day5 of administration are to be calculated by dose.
AUC0-t: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Z-215 | 4 weeks
  Summary statistics of pharmacokinetic parameters on Day1 and Day5 of administration are to be calculated by dose.
AUC0-24: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 hour for Z-215 | 4 weeks
  Summary statistics of pharmacokinetic parameters on Day1 and Day5 of administration are to be calculated by dose.
AUC0-∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Z-215 | 4 weeks
  Summary statistics of pharmacokinetic parameters on Day1 and Day5 of administration are to be calculated by dose.
CL/F: Apparent Total Body Clearance (CL/F) Pharmacokinetic Parameter for Z-215 | 4 weeks
  Summary statistics of pharmacokinetic parameters on Day1 and Day5 of administration are to be calculated by dose.
Vd/F: Apparent Volume of Distribution (Vd/F) Pharmacokinetic Parameter for Z-215 | 4 weeks
  Summary statistics of pharmacokinetic parameters on Day1 and Day5 of administration are to be calculated by dose.
MRT0-∞: Mean Residence Time from Time 0 to Infinity for Z-215 | 4 weeks
  Summary statistics of pharmacokinetic parameters on Day1 and Day5 of administration are to be calculated by dose.
Rac(Cmax): Accumulation Index of Cmax (Rac(Cmax)) for Z-215 | 4 weeks
  Summary statistics of pharmacokinetic parameters on Day1 and Day5 of administration are to be calculated by dose.
Rac(AUC): Accumulation Index of AUC (Rac(AUC)) for Z-215 | 4 weeks
  Summary statistics of pharmacokinetic parameters on Day1 and Day5 of administration are to be calculated by dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan